CLINICAL TRIAL: NCT01974102
Title: Preventing Childhood Obesity Through a Family-Based Mindfulness Intervention
Brief Title: Family Based Mindfulness Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1306012264; 5R21AT007708 (NIH)
Record Dates: First submitted 2013-10-27; First posted 2013-11-01 (Estimated); Results first posted 2021-04-06 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-03

CONDITIONS: Parental Stress; Parent and Child Stress; Parental and Child Obesity; Child Obesity
MeSH Terms: conditions — Pediatric Obesity | interventions — Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- lifestyle (Active Comparator): Attentional control group will receive weekly meeting to view relaxing video and facilitate discussion along with counseling on nutrition and physical activity for 8 weeks.
  Interventions: Behavioral: Lifestyle counseling
- therapy (Experimental): Active group will receive weekly mindfulness based parenting stress reduction (PMH) plus nutrition and physical activity counseling for 8 weeks.
  Interventions: Behavioral: Lifestyle counseling; Behavioral: Parenting Mindfully for Health (PMH)

INTERVENTIONS:
Behavioral: Lifestyle counseling — Active control group will receive weekly session for viewing relaxing video and discussion plus nutritional and physical activity counseling for 8 weeks.
Behavioral: Parenting Mindfully for Health (PMH) — Active participants will receive 8 weeks of mindfulness based parenting stress reduction (PMH) plus nutritional and physical activity counseling for 8 weeks.
  Arms: therapy

SUMMARY:
The goal of the proposed interdisciplinary study is to assess feasibility of recruiting a pilot sample of parents of toddlers and engaging them in a pilot study to test a version of mindfulness-based intervention for parenting stress reduction (PMH), an empirically-supported stress-reduction intervention, plus nutrition and physical activity counseling for parents of preschoolers (aged 2-5); to reduce parent (and child) stress levels; improve parenting; promote healthy eating and physical activity in parent and child; and prevent overweight and obesity in preschoolers with an obese parent.

DETAILED DESCRIPTION:
This project was a preliminary feasibility and pilot efficacy study to assess stressed low income parents of toddlers who were obese to assess whether a mindfulness based parenting intervention (PMH) can reduce their stress, increase parenting and improve family healthy food and physical activity choices. Parents and toddlers also participated in a Toy Wait Task, a behavioral assay of parenting.The empirically-supported stress-reduction intervention, plus nutrition and physical activity counseling (Control) for parents of preschoolers (aged 2-5) was compared to a nutrition and physical activity counseling alone condition to assess whether PMH improved toddler weight, physical activity and parent emotion regulation and healthy eating.

ELIGIBILITY:
Inclusion Criteria:

1. Between ages 18-70 years;
2. Able to read and write (parent)
3. Family with a child between 2-5 years old
4. BMI of parent in obese category
5. High parenting stress (mean score of >=3 on 3 questions from Parenting Stress Index)

Exclusion Criteria:

1. Any psychotic disorder or current psychiatric symptoms for child or parent requiring specific attention, including active symptoms of psychosis or suicidal/homicidal ideation
2. Diagnosis of mental retardation, autism or other pervasive developmental disorder for child
3. Inability to give informed consent
4. Current serious medical disorder precluding participation in physical activity

Ages: 2 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2013-10; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rajita Sinha, PhD, Principal Investigator — Yale University
Locations (1):
- Yale Stress Center, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jastreboff AM, Chaplin TM, Finnie S, Savoye M, Stults-Kolehmainen M, Silverman WK, Sinha R. Preventing Childhood Obesity Through a Mindfulness-Based Parent Stress Intervention: A Randomized Pilot Study. J Pediatr. 2018 Nov;202:136-142.e1. doi: 10.1016/j.jpeds.2018.07.011. Epub 2018 Sep 18. PMID 30241766

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In Phase 1, 20 parent-child dyads started assessments,17 continued post baseline and provided feedback for initial pilot/development phase of PMH+N and C+N interventions. In Phase 2, forty-two parent-preschooler dyads were randomly assigned to receive either the 8-week PMH+N or C+N intervention. Thirty-eight dyads started the intervention
Groups:
- Lifestyle: Both active and control groups will receive counseling on nutrition and physical activity.
  Lifestyle counseling: Active and control participants will receive nutritional and physical activity counseling.
- Prevention Intervention: Active group will receive 8 weeks of mindfulness based parenting stress intervention
  Lifestyle counseling: Active and control participants will receive nutritional and physical activity counseling.
  Mindfulness Based Intervention: Active participants will receive 8 weeks of Mindfulness Based Parenting Stress Intervention
Period: Overall Study
Arm/Group | Lifestyle | Prevention Intervention
Started | 22 | 20
Completed | 15 | 19
Not Completed | 7 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lifestyle | Prevention Intervention | Total
Number analyzed (Participants) | 22 | 20 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] — Age in years via self report
  years
    Age | 31.6 (6.9) | 30.2 (6.3) | 31 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 20 | 42
  Male | 0 | 0 | 0
Race & Ethnicity [Count of Participants; unit: Participants]
  African American, Hispanic and Other | 12 | 14 | 26
  Caucasian | 10 | 6 | 16

OUTCOME MEASURES:

1. Primary Outcome: Attendance
Description: Attendance rates (average number of sessions) were compared across groups.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: Sessions
Groups:
- Lifestyle: Session attendance in Control group
- Prevention Intervention: Session Attendance in Mindfulness based Intervention group
Arm/Group | Lifestyle | Prevention Intervention
Number analyzed (Participants) | 15 | 19
Sessions | 5.7 (1.7) | 7.1 (1.2)
Statistical Analysis 1: Comparison: Lifestyle vs Prevention Intervention; Test type: Superiority; p < 0.015, t-test, 2 sided

2. Secondary Outcome: Change in BMI Percentile
Description: A comparison between groups to determine the impact of the intervention on BMI percentile.
Time Frame: 8 weeks
Population: Children were assessed Pre and Post intervention for weight and height to determine BMI percentiles
Measure: Mean (Standard Deviation); unit: BMI percentile change
Groups:
- Lifestyle: Change in Child BMI Percentile from Post- to Pre- treatment in Control group
- Prevention Intervention: Change in Child BMI Percentile from Post- to Pre- treatment in Mindfulness based Intervention group
Arm/Group | Lifestyle | Prevention Intervention
Number analyzed (Participants) | 15 | 19
BMI percentile change | 12 (25.5) | 1.1 (16.1)
Statistical Analysis 1: Comparison: Lifestyle vs Prevention Intervention; Test type: Superiority; p < 0.03, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 8 weeks
Description: Not different than clinicaltrials.gov definitions
Groups:
- Lifestyle: This group will receive attendance control weekly with attendance in a group to watch a relaxing video and generate discussion.
  Lifestyle counseling: Weekly nutritional and physical activity counseling.
- Prevention Intervention: Active group will receive 8 weeks of parenting mindfully for health (PMH) plus nutrition and physical activity (N) counseling
  Lifestyle counseling: weekly Nutritional and physical activity counseling.
  Mindfulness Based Parenting Intervention: Active participants will receive 8 weeks of Mindfulness Based Parenting Stress Intervention.
Arm/Group | Lifestyle | Prevention Intervention
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/19
Other Adverse Events (participants affected / at risk) | 0/15 | 0/19

LIMITATIONS AND CAVEATS:
Limitations of this study include the small sample size, limited data on the mothers due to participants' time restraints and preference, and short intervention duration.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes